CLINICAL TRIAL: NCT06476392
Title: Melatonin for CHronic BAck Pain (The MOCHA Trial): a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Melatonin for CHronic BAck Pain (The MOCHA Trial)
Acronym: MOCHA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); T&W Engineering A/S (Industry); University of Aarhus (Other); Region of Southern Denmark (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-503530-41-00
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Back Pain Lower Back Chronic; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participating patients, investigators, outcome assessors and statistical analysts are all blinded to treatment allocation. All patient reported data will be filled in by the patient via an online questionnaire using REDCap. An assessor blinded to study treatment will perform all protocol specific objective outcome assessments at baseline and 6 weeks follow-up. Unblinding will first take place after the primary analysis of the data has taken place. A data manager, otherwise, not involved in the study, will prepare the randomization list, using a computerized algorithm in REDCap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): 2 Melatonin tablets (each 5 mg) once daily (egual 10 mg/day) in the evening, 30 min. before going to sleep for 6 weeks. If a participant experiences an adverse event deemed related to the study medication of grade 2 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 the dose will be reduced to 5 mg/day.
  Interventions: Drug: Melatonin 10 MG
- Placebo (Placebo Comparator): 2 identical appearing placebo tablets once daily in the evening, 30 min. before going to sleep for 6 weeks. If a participant experiences an adverse event deemed related to the study medication of grade 2 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 the dose will be reduced to 1 tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 10 MG — 2 Melatonin tablets (each 5 mg) once daily (egual 10 mg/day) in the evening, 30 min. before going to sleep for 6 weeks. If a participant experiences an adverse event deemed related to the study medication of grade 2 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 the dose will be reduced to 5 mg/day.
  Other Names: Melatonin
  Arms: Melatonin
Drug: Placebo — 2 placebo tablets once daily in the evening, 30 min. before going to sleep for 6 weeks. If a participant experiences an adverse event deemed related to the study medication of grade 2 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 the dose will be reduced to 1 tablet.
  Arms: Placebo

SUMMARY:
According to the World Health Organization (WHO) Global Burden of Disease study, back pain is one of the conditions impacting disability the most worldwide.Pain medication use in patients with chronic back pain is substantial, but the efficacy of commonly used analgesics such as paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), muscle relaxants and opioids compared with placebo are modest, with effects typically less than 10 points on a 0-100 pain scale. Importantly, these analgesics are not harmless due to gastrointestinal and cardiovascular side-effects (NSAIDs) and risk of dependency and addiction (opioids). This often leave general practitioners without good treatment options for many patients with chronic low back pain.

More than half of patients with chronic back pain also have sleep problems (i.e. insomnia), which negatively affect daily function, general health and quality of life. Research suggest that insomnia has negative effects on pain processing, and although the relationship between pain and insomnia is bi-directional, insomnia is considered to be a stronger predictor of pain than pain for the development of insomnia.

Melatonin is a widely available drug worldwide, and well known for its use in people with sleep disorders and jetlag. Melatonin is a naturally occurring hormone excreted by the pineal gland that is part of regulating the circadian rhythm (sleep-wake patterns). Unlike commonly used drugs to treat back pain, the safety profile of melatonin is favorable with no adverse events of major clinical significance reported in the treatment of sleep disorders. In recent years, some preliminary studies have showed a promising effect of Melatonin for treatments of pain. A meta-analysis reported an effect size of 0.65 (95%CI 0.34 to 0.96) of Melatonin (doses ranging between 3-10 mg before sleep) compared with placebo in reducing pain in patients with non-musculoskeletal chronic pain (e.g. migraine, irritable bowel syndrome, burning mouth syndrome), suggesting that Melatonin could potentially also be a valid treatment option for chronic musculoskeletal pain patients.

DETAILED DESCRIPTION:
The aim of this randomized double-blind placebo controlled clinical superiority trial is to investigate if daily treatment with Melatonin 10 mg once daily before bedtime for 6 weeks is superior compared with placebo in improving pain intensity assessed at 6 weeks after treatment initiation in patients with chronic back pain.

The primary objective is to compare the effect of the drug Melatonin, relative to placebo, on difference in change in pain intensity (i.e. average pain intensity past 7 days) measured on a 0-10 NRS scale, from baseline to 6 weeks in patients with chronic back pain.

Secondary objectives are to compare the effect of the drug Melatonin, relative to placebo, on 1) pain-related disability, 2) Global Perceived Effect (GPE), 3) insomnia severity, and 4) health-related quality of life. Furthermore, pain trajectory (0 to 6 weeks) and responder indices from baseline to 6 weeks will be compared between the treatment groups for the primary outcome.

Explorative objectives are to investigate changes in pain sensitivity (i.e. pressure pain threshold) and objective sleep metrics as well as effect-modification of presence/absence of comorbid insomnia.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the trial patients must fulfill all the following inclusion criteria:

* Age 18 to 64 years
* Understand and write Danish
* Back pain for 3 months or longer
* Back pain must be present on 'most days' or 'every day' within the past 3 months (will be checked by the question: 'In the past 3 months, how often did you have back pain? - response options: 'never'; 'some days'; 'most days'; 'every day')
* Back pain must limit life or work activities on 'some days', 'most days', or 'every day' within the past 3 months. (will be checked by the question: 'In the past 3 months, how often did your back pain limit your life or work activities? - response options: 'never'; 'some days'; 'most days'; 'every day')
* Average pain intensity of 4 or higher on 0-10 Numeric Rating Scale [NRS] in the past 7 days (ranging from 'no pain' to 'worst imaginable pain').
* All fertile women must use safe contraception (Spiral, birth control pills, contraceptive patch, contraceptive vaginal ring or gestagen injections) for 3 weeks before and 1 week after the trial. If the participants' normal lifestyle includes sexual abstinence, they do not have to use contraception. Instead, they can give an oral informed consent, that they will be sexually abstinent during the trial. A woman is considered non-fertile if she is sterilized, hysterectomized, bilateral oophorectomized or is postmenopausal. A woman is considered postmenopausal when vaginal bleeding has been absent for 1 year (reported by the participant).

Exclusion Criteria:

Patients will be excluded based on any of the following exclusion criteria:

* Known abuse of alcohol or other substances
* Self-selected non-user of e-boks
* Opioid use (reported by participant)
* Known malignancies within past 6 months (reported by participant)
* Known fractures within past 4 months (reported by participant)
* Known lumbar radiculopathy (reported by participant)
* Known spinal stenosis (reported by participant)
* Severe psychiatric disorders and/or psychotic symptoms evaluated by the investigator (reported by participant)
* Suicide and self-damage thoughts (reported by participant)
* Inflammatory/autoimmune arthritis (reported by participant)

Patients with contraindications to Melatonin according to the Danish Medicines Agencys approved product information:

* Moderate to severe kidney insufficiency (GFR < 30 mL/min)
* Moderate to severe liver insufficiency (ALAT must not be elevated more than 3-fold over highest reference level)
* Auto-immune diseases
* Epilepsy
* Warfarin use
* Benzodiazipin use (including hypnotics)
* Fluvoxamin use (Ciprofloxacin, Norfloxacin)
* Calcium antagonist use (Verapamil, Nifedepin)
* Pregnancy or pregnancy-wish or breastfeeding (a negative pregnancy test has to be available for all fertile female patients at baseline)
* Intolerance to melatonin

For the EEG subgroup:

If the anatomy of the outer ear making it impossible to do ear EEG monitoring If there have a perforation of the tympanic membrane (eardrum) If they have an ear tube in the tympanic membrane If their ear piercings that are not compatible with ear EEG. If they use anticoagulants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change in average pain intensity during the last 7 days between groups | Difference in change from baseline to 6 weeks
  Average pain intensity during last 7 days will be assessed on a 0-10 Numeric Rating Scale (NRS) (ranging from 'no pain to 'worst imaginable pain')

SECONDARY OUTCOMES:
Insomnia severity | Baseline and after 6 weeks
  Insomnia will be assessed with the Insomnia Severity Index (ISI), which is a brief 7 item patient-reported instrument with a score ranging from 0-28 (0=best;28=worst)
Weekly pain intensity score trajectory | Weekly from baseline to 6 weeks
  The trajectory of weekly numerical rating scale (NRS) pain intensity scores assessed on a 0-10 Numeric Rating Scale (NRS) (ranging from 'no pain to 'worst imaginable pain') from baseline to 6 weeks
30% pain intensity responders | Change from baseline to 6 weeks
  Difference in number of patients with more than 30% improvement in pain intensity from baseline to 6 weeks
50% pain intensity responders | Change from baseline to 6 weeks
  Difference in number of patients with more than 50% improvement in pain intensity from baseline to 6 weeks
Global Perceived Effect (GPE) for pain | After 6 weeks
  Assessment of overall change in pain from baseline to 6 weeks. Participants will be asked at 6 weeks: 'How is your pain now compared to when you entered this study', with 5 response options (much worse, worse, almost the same/unchanged, improved, much improved)
Physical and Mental Health | Baseline and after 6 weeks
  Physical and Mental Health will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS-10) Global Health questionnaire version 1.2. Difference in change in physical and mental health scores between treatment groups from baseline to 6 weeks. PROMIS-10 consist of 10 questions concerning different aspects of global health. The first 9 questions are score on a Likert scale with 5 response options, and the last question asks about pain using a 0-10 numeric rating scale
Back pain related disability | Baseline and after 6 weeks
  Back pain related disability will be assessed using the Roland Morris Disability Questionnaire (RMQ). RMQ is a 23-item questionnaire (RMQ) developed to assess functional limitation and disability among patients with low back pain. The RMQ 23-item version will be used because 1) it has been cross-culturally validated in Danish (the original RMQ 24-item version has not), 2) the psychometric properties of the 23 vs 24 item RMQ have been shown to be similar. Each of the 23 items is yes/no (scored as 1 and 0 points respectively) with the scale ranging from 0 (no disability) to 23 (extremely severe disability).

OTHER OUTCOMES:
Time from sleep onset until final awakening (TST) from Ear EEG in subgroup of 60 patients | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Sleep efficiency (SE) from Ear EEG in subgroup of 60 patients | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM). SE is the ratio of TST to time in bed / 100%
Sleep onset latency (SOL) from Ear EEG in subgroup of 60 patients | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Wake after sleep onset (WASO) from Ear EEG in subgroup of 60 patients | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
REM sleep latency from Ear EEG in subgroup of 60 patients | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Time from sleep onset until first epoch of REM stage sleep from Ear EEG | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Amount of wake and stage N1, N2, N3, and R sleep as a percentage of SPT from Ear EEG | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Number of awakenings within TST from Ear EEG | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Arousal index which is number of arousals per hour from Ear EEG | Baseline and week 4.
  Difference in change in sleep metric between treatment groups (Melatonin [n=30] vs.placebo [n=30]) from baseline to 4 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Ease-of-use and Comfort with ear EEG | Baseline and week 4.
  Three 0-10 questions are used: 1) How did you experience falling asleep with the ear EEG device, 2) How did you experience sleeping with the ear EEG device?, 3) How would you rate your experience of soreness or discomfort in your ears after sleeping with the device? A lower sum score is worse.
Ear EEG adverse device effects | Baseline and week 4.
  Any adverse device effect defined as an adverse effect related to the use of the ear EEG
Age | Baseline
  The age of the participant will be calculated using the date of randomisation and the date of birth.
Sex | Baseline
  The sex of the participant assigned at birth (male or female)
Height | Baseline
  Self-reported in centimeter
Weight | Baseline
  Self-reported in kilograms
Marital status | Baseline
  Self-reported marital status
Level of education | Baseline
  The categories for level of education are compulsory education, upper secondary, bachelor degree, master degree, Phd degree
Concomitant medication | Baseline
  Self-reported concomitant medication will be recorded in the eCRF by a trained nurse during the information visit.
Medical history and concomitant illnesses | Baseline
  Self-reported medical history and concomitant illnesses relevant to the investigation will be recorded in the eCRF. A clinically significant worsening of a concomitant illness will be reported as an AE
Blood pressure | Baseline
  Diastolic and systolic
Heart rate | Baseline
  Beats per min
Serum levels of Alanintransaminase (ALAT) | Baseline
  Blood test
Serum levels of creatinine | Baseline
  Blood test
Serum levels of Glomerular Filtration Rate (GFR) | Baseline
  Blood test
Choriogonadotropin (hCG) | Baseline and week 3
  Urine test for pregnancy
Pain sensitivity | Baseline and after 6 weeks.
  Pressure pain threshold is assessed using a handheld algometer. Pressure pain thresholds will be assessed locally at the right erector spinae muscle (3 cm from the fourth lumbar spinous process) and at the left upper trapezius muscle (10 cm horizontally from the acromion in direct line with the seventh cervical spinous process).
Smoking status | Baseline
  Self-reported
Alcohol consumption | Baseline
  Self-reported
Physical activity level | Baseline
  Self-reported
Work status | Baseline
  Self-reported
Chronic pain | Screening
  Chronic pain will be assessed using the Graded Chronic Pain Scale Revised (GCPS-R) questionnaire. The GCPS-R is a brief, freely available questionnaire that assesses frequency and severity of pain and its impact. The GCPS-R uses 5 items to categorize pain into no chronic pain, mild chronic pain, bothersome chronic pain, and high-impact chronic pain
Harms | Week 3, week 6 and week 8
  In both groups the following will be reported:
  Number of deaths Number of SAE Number of AE and categorized in mild and moderate

CONTACTS AND LOCATIONS:
Overall Officials: Karin Due Bruun, PhD, Principal Investigator — University Hospital Odense
Locations (1):
- Pain Center, University Hospital Odense, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilic K, Vaegter HB, Bruun KD, Vach W, Hartvigsen J, Koes BW, Kidmose P, Sondergaard J, Thorlund JB. Melatonin for chronic back pain (the MOCHA trial): study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2025 Nov 17;26(1):513. doi: 10.1186/s13063-025-09206-w. PMID 41250112